CLINICAL TRIAL: NCT04140201
Title: Evaluation of Lipid Lowering Agents on Diabetic Retinopathy and Cardiovascular Risk of Diabetic Patients
Brief Title: Effect of Lipid Lowering Agents on Diabetic Retinopathy and Cardiovascular Risk of Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alaa Hassan ElBaz (Other)
Responsible Party: Sponsor-Investigator, Alaa Hassan ElBaz, Assistant lecturer at beni suef university, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diabetic Retinopathy
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Fenofibrate; Fibric Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Receive oral hypoglycemic +omega 3 (Active Comparator): Eicosapentanoic acid + standard treatment
  Interventions: Drug: Omega 3 fatty acid
- Receive oral hypoglycemic +statin (Active Comparator): Simvastatin + standard treatment
  Interventions: Drug: Simvastatin 40mg
- Receive oral hypoglycemic +fibrate (Active Comparator): Fenofibrate +standard treatment
  Interventions: Drug: Fenofibrate 200mg
- Receive oral hypoglycemic only (No Intervention): Standard treatment only

INTERVENTIONS:
Drug: Simvastatin 40mg — Drugs that lower lipid level
  Other Names: Statin
  Arms: Receive oral hypoglycemic +statin
Drug: Fenofibrate 200mg — Drugs that lower lipid levels
  Other Names: Fibrate
  Arms: Receive oral hypoglycemic +fibrate
Drug: Omega 3 fatty acid — Drugs that lower lipid levels
  Other Names: n3 FA
  Arms: Receive oral hypoglycemic +omega 3

SUMMARY:
The investigator study evaluate the effect of different lipid lowering agents on the progression of diabetic retinopathy and other reduction of cardiovascular risk of diabetic patients

DETAILED DESCRIPTION:
The investigator study compare the effect of lipid lowering agent on the enhancement of visual acuity and on reduction of macular edema in patients with diabetic retinopathy and also compare their effect on reduction of cardiovascular risk on diabetic patients via assessment of ASCVD risk score

ELIGIBILITY:
Inclusion Criteria:

* type 2diabetes
* Non proliferative diabetic retinopathy

Exclusion Criteria:

* Uncontrolled glycemic level
* proliferative diabetic retinopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The 80 participants will be evaluated through reduction of macular edema | 18 weeks
  assessed by ocular coherence tomography

SECONDARY OUTCOMES:
The 80 participants will be evaluated through reduction of cardiovascular risk | 18 weeks
  assessed by ASCVD risk score